CLINICAL TRIAL: NCT02449031
Title: A Prospective Observational Study in Cystic Fibrosis Patients With Chronic Respiratory Pseudomonas Aeruginosa Infection Treated With TOBI® PODHALER® (Tobramycin Inhalation Powder) or Other FDA Approved Inhaled Antipseudomonal Antibacterial Drugs
Brief Title: Observational Study in Cystic Fibrosis Patients Using TOBI® PODHALER® or Other FDA Approved Inhaled Antipseudomonal Antibacterial Drugs
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: CTBM100C2407
Record Dates: First submitted 2015-05-04; First posted 2015-05-20 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Pseudomonas Aeruginosa in Cystic Fibrosis
MeSH Terms: interventions — Tobramycin; Aztreonam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TOBI® PODHALER® cohort
  Interventions: Drug: TOBI® PODHALER®
- non-TOBI® PODHALER® cohort: Approximately 250 patients treated with other FDA-approved inhaled antipseudomonal antibacterial drugs at enrollment
  Interventions: Drug: TOBI®; Drug: Bethkis®; Drug: Cayston®

INTERVENTIONS:
Drug: TOBI® PODHALER®
  Groups: TOBI® PODHALER® cohort
Drug: TOBI® — tobramycin inhalation solution, USP
  Groups: non-TOBI® PODHALER® cohort
Drug: Bethkis® — tobramycin inhalation solution
  Groups: non-TOBI® PODHALER® cohort
Drug: Cayston® — aztreonam for inhalation solution
  Groups: non-TOBI® PODHALER® cohort

SUMMARY:
This is a multicenter, prospective, two cohort, observational study over a 5-year period in Cystic Fibrosis (CF) patients with chronic Pseudomonas aeruginosa infection.The study will collect data over 1 year on respiratory function, antibacterial effectiveness, and clinical outcomes of treatment with inhaled antipseudomonal antibiotics and data over 5 years on microbiological and safety assessments.

DETAILED DESCRIPTION:
This study will include CF patients chronically colonized with P. aeruginosa enrolled in the Cystic Fibrosis Foundation (CFF) PortCF registry and using TOBI® PODHALER® or another FDA-approved inhaled antipseudomonal antibiotic. No therapeutic intervention will be assigned and physicians will use their discretion in choosing a treatment regimen for their patients.

Sputum samples (primarily collected during routine clinical follow-up) from patients able to spontaneously produce sputum will be sent to a central laboratory for analysis.

In addition, this study will include two optional sub-studies for qualifying patients in the first study year - Sputum microbiology sub-study and TOBI® PODHALER® sputum pharmacokinetics (PK) sub-study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 years of age.
* Documented FEV1 ≥ 25% predicted in the previous year.
* Diagnosis of cystic fibrosis.
* Established diagnosis of chronic P. aeruginosa infection of the lungs defined as two or more positive P. aeruginosa cultures in the previous year as documented in the subject's medical history (this may include a history of one positive culture in the year prior to enrollment and one positive culture from the specimen collected at the baseline visit).
* Prescribed and initiated chronic treatment with FDA-approved inhaled antipseudomonal antibiotic for chronic P. aeruginosa infection (e.g. TOBI® PODHALER®, TOBI®, Cayston® and Bethkis®).
* Actively enrolled or willingness to enroll in PortCF registry.
* Willing and able to provide written informed consent or, parent/guardian consent and where applicable pediatric assent, for participation and use of relevant clinical data previously captured in PortCF.
* Anticipated to have good adherence to routine visits, defined as the investigator having good knowledge that the patient has been to at least 2-3 routine visits in the previous year.

Exclusion Criteria:

* Documented FEV1 < 25% predicted in the previous year.
* Current participation in an interventional clinical study with an inhaled antibiotic treatment.
* Treatment with compounded tobramycin (e.g. the use of tobramycin IV solution adapted for use by inhalation).
* Treatment with inhaled antipseudomonal antibacterial drug(s) that are not FDA approved.
* Patients undergoing an early eradication regimen for CF (first line therapy).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients chronically colonized with P. aeruginosa enrolled in the Cystic Fibrosis Foundation (CFF) PortCF registry and using TOBI® PODHALER® (TOBI® PODHALER®-treated cohort) or another FDA-approved inhaled antipseudomonal antibiotic (non-TOBI® PODHALER®-treated cohort).
  It is anticipated that this patient population will include a subset of patients with increased P. aeruginosa MICs to tobramycin at baseline.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Absolute change in forced expiratory volume in one second (FEV1) percent predicted from baseline. | 1 year
Absolute change from baseline in the number of P. aeruginosa colony forming units in sputum. | 1 year
Minimum inhibitory concentration (MIC) of tobramycin and the following antipseudomonal antibacterial drugs (meropenem, imipenem, ceftazidime, aztreonam and ciprofloxacin) for P. aeruginosa sputum isolates in both treatment cohorts. | Up to 5 years
Frequency of the following treatment emergent pathogens in sputum: S. aureus (MRSA and MSSA), S. maltophilia, A. xylosoxidans, and Burkholderia spp.in both treatment cohorts. | Up to 5 years
Number of pulmonary exacerbations and those leading to hospitalization. | 1 year
Proportion of patients experiencing pulmonary exacerbations including those leading to hospitalization. | 1 year
Incidence rate of patients with one or more pulmonary exacerbations. | 1 year
Incidence rate of pulmonary exacerbations. | 1 year
Time to first pulmonary exacerbation. | 1 year
Use of additional antipseudomonal antibiotics (overall, IV, oral) to treat pulmonary exacerbations. | 1 year
Mortality rate | 1 year
Pharmacokinetic properties of TOBI® PODHALER® as measured by sputum specimens collected during the on-treatment cycles. | 1 year
Number of respiratory related hospitalizations. | 1 year
Duration of stay for respiratory related hospitalizations. | 1 year
Number of non-respiratory related hospitalizations. | 1 year
Duration of stay for non-respiratory related hospitalizations. | 1 year

SECONDARY OUTCOMES:
Relative change in FEV1 % predicted from baseline. | 1 year

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Novartis Investigative Site, Anchorage, Alaska
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Bellflower, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Madera, California
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Grand Rapids, Michigan
  - Novartis Investigative Site, Ypsilanti, Michigan
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Billings, Montana
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, New Hyde Park, New York
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Hershey, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Sioux Falls, South Dakota
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Spokane, Washington